CLINICAL TRIAL: NCT07052994
Title: A Phase Ia/Ib Trial of Revumenib Combined With Cytarabine, Daunorubicin, and Gemtuzumab Ozogamicin (GO) in Frontline and Relapsed /Refractory Pediatric Acute Leukemia Patients
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1396; NCI-2025-04739 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-06-30; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Pediatric Acute Leukemia
MeSH Terms: interventions — revumenib; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose Escalation of Revumenib in combination with cytrabine and Daunorubicin and GO (Experimental): Treatment will be administered on an inpatient basis
  Interventions: Drug: Revumenib; Drug: Cytrabine; Drug: Daunorubicin
- Dose Expansion of Revumenib in combination with cytrabine and Daunorubicin and GO (Experimental): Treatment will be administered on an inpatient basis
  Interventions: Drug: Revumenib; Drug: Cytrabine; Drug: Daunorubicin

INTERVENTIONS:
Drug: Revumenib — Given by IV
Drug: Cytrabine — Given by IV
Drug: Daunorubicin — Given by IV

SUMMARY:
The goal of Phase 1a of this clinical research study is to find the highest tolerable dose of revumenib that can be given in combination with cytarabine, daunorubicin, and gemtuzumab ozogamicin to patients who have acute leukemia.

The goal of Phase 1b of this clinical research study is to learn if the dose of revumenib in combination with cytarabine, daunorubicin, and gemtuzumab ozogamicin found in Phase 1a can help to control the disease.

DETAILED DESCRIPTION:
Primary Objective:

To determine the safety, tolerability and recommended phase II dose (RP2D) of Revumenib incombination with cytarabine and daunorubicin and Gemtuzumab ozogamicin (GO) in relapsed refractory and frontline pediatric patients with acute leukemias, with primary endpoint defined as DLT (per Section 7.5)

Secondary Objective:

To determine the preliminary assessment of efficacy by overall response (OR), including complete remission (CR), CR with incomplete blood count recovery and partial remission, overall survival (OS), event-free survival (EFS) and duration of response (DOR) of pediatric patients treated with this combination.

Exploratory Objective:

To evaluate molecular and cellular markers that may be predictive of antitumor activity and/or resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Age . 6 months - 21 years of age.
2. ECOG performance status of < 2.
3. Phase 1a portion of the study: Relapsed/refractory AML, or MPAL per ELN/NCCN with a myeloid phenotype with KMT2Ar, NPM1c, NUP98r and UBTF-ITD.
4. Phase 1b portion of the study: Frontline AML, or MPAL per ELN/NCCN with a myeloid phenotype with KMT2Ar, NUP98r and UBTF-ITD.
5. WBC must be below 25,000/ ƒÊL at time of enrollment. Patients may receive cytoreduction prior to enrollment.
6. Baseline ejection fraction must be > 50%.
7. Adequate hepatic function (direct bilirubin < 2x upper limit of normal (ULN) unless increase is due to Gilbert's disease or leukemic involvement, and AST and/or ALT < 3x ULN unless considered due to leukemic involvement, in which case direct bilirubin or AST and/or ALT < 5x ULN will be considered eligible).
8. Potassium should be maintained at . 4.0 mEq/L and magnesium at > 2.0 mg/dL. Maintenance PO supplementation should be started for patients who are below these thresholds, and Revumenib dosing instructions as provided in Table 2 should be followed.
9. Adequate renal function (creatinine clearance .
10. Willing and able to provide informed consent.
11. The time between the previous treatment and the start of the new treatment will be at least 14 days for both cytotoxic and non-cytotoxic therapies, including immunotherapies, or it will be equivalent to 5 half-lives of the prior therapy, whichever is shorter.
12. Oral hydroxyurea and/or cytarabine (up to 2 g/m2) for patients with rapidly proliferative disease is allowed before the start of study therapy, as needed, for clinical benefit and after discussion with the PI. Concurrent therapy for central nervous system (CNS) prophylaxis or continuation of therapy for controlled CNS disease is permitted.
13. Women of childbearing potential must agree to adequate methods of contraception during the study and at least 4 months (120 days) after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study and at least 4 months (120 days) after the last treatment.

Exclusion Criteria:

1. Patients with any concurrent uncontrolled medical condition, laboratory abnormality, or psychiatric illness which could place the patient at unacceptable risk of study treatment.
2. The use of other chemotherapeutic agents or anti-leukemic agents is not permitted during study with the following exceptions (1) intrathecal chemotherapy for prophylactic use or for controlled CNS leukemia. (2) use of hydroxyurea for patients with rapidly proliferative disease or for control of counts during differentiation syndrome. (3) use of steroids for treatment of differentiation syndrome.
3. Patients with any severe gastrointestinal or metabolic condition which could interfere with the absorption of oral study medications.
4. Patients with a concurrent active malignancy under treatment.
5. Known active hepatitis B (HBV) or Hepatitis C (HCV) infection or known HIV infection.
6. Female subjects who are pregnant or breast-feeding.
7. Patient has an active uncontrolled infection.
8. Any of the following within the 6 months prior to study entry: myocardial infarction, uncontrolled/unstable angina, congestive heart failure (New York Heart Association Classification Class .II), life-threatening, uncontrolled arrhythmia, cerebrovascular accident, or transient ischemic attack.
9. QTc >450 msec for males and QTc >470 msec for females using the Fridericia Formula.
10. History of or any concurrent condition, therapy, or laboratory abnormality that in the Investigator's opinion might confound the results of the study, interfere with the patient fs participation for the full duration of the study, or is not in the best interest of the patient to participate.
11. Clinically active central nervous system (CNS) leukemia.
12. Patients on immunosuppressive therapy post-HSCT at the time of screening with R/R leukemia (must be off all systemic immunosuppression therapy for at least 2 weeks and calcineurin inhibitors for at least 4 weeks). The use of topical steroids for cutaneous graft-versus-host disease (GVHD) or stable systemic steroid doses less than or equal to 0.2-0.3mg/kg of prednisone daily are permitted.
13. Patients GVHD grade >1 is not allowed.

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2032-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Branko Cuglievan, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org